CLINICAL TRIAL: NCT03933007
Title: Comparison of Maximum Blood Concentrations of Colchicine Between Responders and Non-responders to Colchicine Treatment During Gout Flare
Brief Title: Relation Between Blood Concentration of Colchicine and Response to Colchicine Treatment in Gout Flare
Acronym: COMpARE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: faillure of recrutement
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P170409J; 2018-002542-37 (EudraCT Number)
Record Dates: First submitted 2019-02-08; First posted 2019-05-01 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Gout Flare
MeSH Terms: interventions — Colchicine; Midazolam; fexofenadine

STUDY DESIGN:
Intervention Model Description: all participants will perform the pharmacokinetic study and take colchicine 1 mg + 0.5 mg 1 hour later, midazolam 1 mg and fexofenadine 120 mg.
  A pharmacokinetic study is an interventional study with only one arm.
Masking Description: all participants will perform the pharmacokinetic study and take colchicine 1 mg + 0.5 mg 1 hour later, midazolam 1 mg and fexofenadine 120 mg.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pharmacokinetic study (Other): all participants will undergo pharmacokinetic study and take colchicine (1.5 mg over 1 hour), midazolam (1 mg) and fexofenadine (120 mg)
  Interventions: Drug: Colchicine,; Drug: midazolam,; Drug: fexofenadine

INTERVENTIONS:
Drug: Colchicine, — the day of phenotyping assay
  * Colchicine : 1.5 mg over 1 hour (1 mg + 0.5 mg 1 hour later)
Drug: midazolam, — Midazolam 1 mg
Drug: fexofenadine — Fexofenadine 120 mg

SUMMARY:
Gout, secondary to sodium urate crystal deposition, is responsible of recurrent inflammatory painful flares. Efficacy of colchicine which is the first line drug for the treatment and prophylaxis of gout flare varies and only half of treated patients experience good response. This study aims to optimize colchicine prescription for the treatment and prophylaxis of gout flare.

Current data suggest that efficiency of colchicine relies on its maximum blood concentration (Cmax).

In this study, the investigators hypothesize that responders to colchicine treatment have higher colchicine Cmax than non-responder patients following the recommended dose regimen (1 mg then 0.5 mg 1 hour later).

The individual pharmacokinetics (PK) of colchicine remains poorly investigated while the assessment of individual drug metabolisms can be performed.

The hypothesis of this study stands that several factors contribute to the variability of colchicine Cmax. The analysis of individual PK profile and a well-characterized metabolism of colchicine will permit a personalized treatment regimen for the treatment and prophylaxis of gout flares.

DETAILED DESCRIPTION:
Gout flare is driven by interleukin (IL)-1β production and can be treated by colchicine, NSAID, corticoid or IL-1β blockers (PMID 27457514).

Colchicine is an alkaloid compound that disrupts cytoskeletal functions through inhibition of microtubule polymerization and consequently interferes with the intracellular assembly of the inflammasome NLRP3 complex that mediates activation of IL-1β (PMID 16407889).

Efficacy of colchicine treatment in gout flare varies between 37.5 and 64% (PMID 3314832; 20131255). Previous study suggests that colchicine efficiency relies on its blood maximum concentration (Cmax) (PMID 20131255). However this hypothesis needs to be confirmed.

The hypothesis of this study stands that colchicine Cmax varies with individual colchicine pharmacokinetics and that this individual variation may explain the variation response of colchicine treatment.

Absorption of orally administrated colchicine varies between 24 et 88% with an average of 45%. Thus, following oral administration of 1.8 mg colchicine over 1 hour to healthy young adults, under fasting condition, the colchicine Cmax (mean 6.2 ng/ml) is reached within a median of 1.8 hours (range 1.0-2.5) (PMID 20131255).

Colchicine is demethylated to two metabolites, 2-O-demethylcolchicine and 3-O-demethylcolchicine (2- and 3-DMC, respectively). In vitro studies have shown that hepatic cytochrome P450 3A4 (CYP3A4) is involved in the metabolism of colchicine to 2- and 3-DMC. Colchicine is also a substrate of liver and intestinal P-glycoprotein (P-gp) transporter.

Colchicine is eliminated in urine and stools. 40-65% of orally administrated colchicine is recovered unchanged in urine. Enterohepatic recirculation and biliary excretion account for around 50% of colchicine elimination. The mean half-live elimination is 20 to 40 hours.

Thus, blood concentration of colchicine depends on kidney and hepatic functions, intestinal absorption and secretion, the presence of drug-drug interactions and individual characteristics of CYP3A4 and P-gp activities (PMID 21480191).

The individual CYP3A4 and P-gp activities can be assessed with specific probe and/or substrate of these proteins in the so-called phenotyping assay. Thus, using micro dose of midazolam and fexofenadine the activity of CYP3A4 and P-gp, respectively, can be determined and subsequently the individual pharmacokinetic profile of colchicine characterized (PMID 24722393).

CYP3A4 activity is given by the ratio of hydroxy-midazolam/midazolam assessed 2 hours after an oral administration of 1 mg midazolam (PMID 24722393).

P-gp activity is given by the area under the curve (AUC) of a short kinetic that measures fexofenadine concentrations at 2, 3 and 6 hours after its oral administration of 120 mg (PMID 24722393).

These CYP3A4 and P-gp activities will be correlated with blood colchicine concentrations determined at different time points after an oral administration of 1.5 mg over 1 hour under fasting condition.

The CYP3A4 and P-gp phenotyping will be proposed to all gouty patients who experienced gout flare and who fulfilled the inclusion and exclusion criteria.

Participants will have 3 visits :

* V0: inclusion visit of patients who had untreated gout flare. Signed consent to the study will be collected and blood analysis performed. A blood collection and biobank of serum will be done using the blood harvested for gout care. Colchicine will be initiated at 1.5 mg over 1 hour (1 mg + 0.5 mg)
* V1: treatment efficiency will be assessed 48 h after V0 using Visual Analogue Scale (VAS) (0-100) pain measurement. Patients who will have an improvement of VAS more than 50% of baseline VAS will be considered as responders to colchicine. In contrast an improvement less than 50% of baseline VAS will be considered as non-responders. Gout flare treatment will be adapted according to patient response. Colchicine treatment will be stopped after gout flare resolution
* V2: this visit will be appointed 1 month after V1 (far enough after resolution of gout flare). During this visit, the CYP3A4 and P-gp phenotyping will be performed. Patients will receive colchicine (1.5 mg over 1 hour) and midazolam (1 mg) and fexofenadine (120 mg) orally. A kinetic of blood samples will be harvested with a total of 8 time points from T0 prior to drug administration to T6 6 hour post-drug administration. At the end of the phenotyping kinetic, urate-lowering therapy will be introduced according to usual care and dosage. This visit is the last visit of the protocol and patients will be followed-up as usual care.

Plasma concentrations of colchicine, midazolam, hydroxymidazolam and fexofenadine will be quantified by liquid chromatography-tandem mass spectrometry (PMID 24295116).

Plasma concentrations of colchicine will then correlate to CYP3A4 and P-gp activities estimated by midazolam and fexofenadine metabolism, respectively.

The phenotyping will be performed in 34 colchicine responder and 34 colchicine non-responder patients.

ELIGIBILITY:
Inclusion Criteria:

Patients (> 18 years old) with gout flare defined by following items :

* Identification of sodium urate crystals in synovial fluid analysis
* Or gout flare diagnosis according to Nijmegen criteria (score > 8/13)

  * Man (2 pts)
  * History of flare (2 pts)
  * Flare involving first metatarsophalangeal joint (2.5 pts)
  * Maximum of flare within 24h (0.5pt),
  * Redness (1 pt),
  * History of hypertension or cardiovascular diseases (1.5 pts),
  * Serum urate level > 360 µmol/l during flare (3.5 pts)
* Duration of flare < 48 h
* Monoarticular involvement

Exclusion Criteria:

* Hypersensitivity to colchicine, fexofenadine, benzodiazepine or the excipients of these drugs
* Contra-indication to colchicine : chronic kidney disease stage 4-5, severe hepatic impairment, treatment by macrolide antibiotics
* Used of pain-killers other than acetaminophen
* Involvement in another clinical trial with drug administration
* Illiteracy
* Pregnant woman or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration of colchicine | From drug administration to 6 hour post-drug administration
  Maximum plasma concentration of colchicine in responders and non-responders to colchicine treatment for gout flare during pharmacokinetic study performed 1 month after flare resolution and before initiation of urate-lowering therapy.

SECONDARY OUTCOMES:
Maximum Plasma Concentration [Cmax] | From drug administration to 6 hour post-drug administration
  pharmacokinetic parameter of absorption of colchicine
Time needed to reach Cmax [Tmax ] | From drug administration to 6 hour post-drug administration
  pharmacokinetic parameter of absorption of colchicine
Absorption rate constant [Ka] | From drug administration to 6 hour post-drug administration
  pharmacokinetic parameter of absorption of colchicine
Volume of distribution [Vd] | From drug administration to 6 hour post-drug administration
  pharmacokinetic parameter of distribution of colchicine
Area under the curve [AUC] | From drug administration to 6 hour post-drug administration
  pharmacokinetic parameter of distribution of colchicine
Clearance | From drug administration to 6 hour post-drug administration
  pharmacokinetic parameter of elimination of colchicine

CONTACTS AND LOCATIONS:
Overall Officials: Hang-Korng EA, PhD, MD, Principal Investigator — AP-HP - Groupe hospitalier Lariboisière Fernand Widal
Locations (1):
- Hôpital Lariboisière-Service de Rhumatolologie, Paris, France